CLINICAL TRIAL: NCT00751101
Title: Pilot Study of Nicotine Patches to Reduce Hand-Foot Syndrome Associated With Capecitabine Chemotherapy in Patients With Metastatic Breast Cancer
Brief Title: Nicotine Patches in Reducing Hand-Foot Syndrome in Patients Who Are Receiving Capecitabine For Metastatic Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low Accrual
Sponsor: University of California, San Francisco (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 057514; ROCHE-UCSF-057514 (Other: University of California, San Francisco); NCI-2011-03236 (Registry Identifier: NCI Clinical Trials Reporting Program (CTRP))
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Breast Cancer; Chemotherapeutic Agent Toxicity; Palmar-plantar Erythrodysesthesia
Keywords: palmar-plantar erythrodysesthesia; chemotherapeutic agent toxicity; stage IV breast cancer; recurrent breast cancer
MeSH Terms: conditions — Breast Neoplasms; Hand-Foot Syndrome | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A: Prior to initiation of capecitabine (Experimental): Patients apply a transdermal nicotine patch once every 24 hours beginning 1 day prior to initiation of capecitabine and continuing until the end of capecitabine therapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nicotine patch
- Arm B: After hand-foot syndrome symptoms appear (Experimental): Patients apply a transdermal nicotine patch once every 24 hours beginning with the course of chemotherapy initiated after hand-foot syndrome symptoms appear and continuing until the end of capecitabine therapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Nicotine patch

INTERVENTIONS:
Drug: Nicotine patch — Nicotine patch applied prior to and concurrently with capecitabine chemotherapy or beginning during the first course of capecitabine after the onset of hand-foot syndrome symptoms

SUMMARY:
RATIONALE: Nicotine patches may reduce hand-foot syndrome in patients receiving capecitabine for metastatic breast cancer. It is not yet known which nicotine patch regimen may be more effective in reducing hand-foot syndrome.

PURPOSE: This randomized clinical trial is studying which schedule of using nicotine patches is more effective in reducing hand-foot syndrome in patients who are receiving capecitabine for metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility of using nicotine patches, in terms of side effects and the number of voluntary withdrawals from the study, in patients with metastatic breast cancer undergoing chemotherapy with capecitabine.

Secondary

* Determine the efficacy of nicotine patches as preventive agents for hand-foot syndrome (HFS) by assessing the incidence of HFS in each arm.
* Determine the grade of HFS in each arm.
* Determine the percentage of patients requiring a reduction in dose of capecitabine due to adverse events.
* Determine the percentage of patients requiring pain medication for HFS.
* Determine the percentage of patients using other symptomatic treatments for HFS (e.g., moisturizers, ice, cooling packs).
* Evaluate the effect of nicotine patches on quality-of-life of patients undergoing capecitabine chemotherapy.

OUTLINE: This is a multicenter study. Patients are randomized to 1 of 2 treatment arms.

Patients receive oral capecitabine twice daily on days 1-7 and 15-21. Treatment with capecitabine repeats every 21 days for up to 5 courses in the absence of disease progression or unacceptable toxicity.

* Arm I: Patients apply a transdermal nicotine patch once every 24 hours beginning on 1 day prior to initiation of capecitabine and continuing until the end of capecitabine therapy in the absence of disease progression or unacceptable toxicity.
* Arm II: Patients apply a transdermal nicotine patch once every 24 hours beginning on day 1 of the course of chemotherapy following the appearance of hand-foot syndrome symptoms. Treatment continues until the end of capecitabine therapy in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, and at 3 and 12 weeks. Patients also complete a daily diary to document side effects and medication compliance.

After completion of study therapy, patients are followed at 3 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Metastatic disease
* Scheduled to begin treatment with capecitabine at the University of California, San Francisco (UCSF) Cancer Center, San Francisco General Hospital, or Cornell Medical Center
* No concurrent hand-foot syndrome (HFS) due to other medications

  * Prior HFS due to other medications allowed provided that the symptoms have been completely resolved for ≥ 4 weeks prior to study entry
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Menopausal status not specified
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* Able to participate in study procedures and quality-of-life evaluations and willing to comply with study requirements
* Non-English speaking patients are allowed provided they demonstrate adequate understanding of the study rationale and procedures and can give voluntary consent with the aid of a translator
* No clinically significant cardiac or peripheral vascular disease or symptom, including any of the following:

  * History of myocardial infarction
  * Congestive heart failure
  * Cardiac arrhythmias (including atrial fibrillation)
  * Cardiac or vascular bypass
  * Uncontrolled hypertension
  * Unstable angina
  * Undiagnosed arrhythmias or claudication
* No Alzheimer disease, Parkinson disease, or active psychiatric disease
* Not currently smoking

  * Patients who are former smokers must have stopped smoking ≥ 6 months prior to study entry
* No known hypersensitivity to nicotine patches

PRIOR CONCURRENT THERAPY:

* At least 6 months since prior and no other concurrent nicotine patches
* Prior chemotherapy allowed, except capecitabine for treatment of metastatic disease
* Concurrent other symptomatic treatment for hand-foot syndrome (HFS) (e.g., usual skin care, topical moisturizers, ice packs, pain medications) allowed
* No concurrent pyridoxine

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-08-20 (Actual); Primary Completion 2014-03-24 (Actual); Study Completion 2018-03-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hope S. Rugo, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B: After Hand-foot Syndrome (HFS) Symptoms Appear: Patients apply a transdermal nicotine patch once every 24 hours beginning with the course of chemotherapy initiated after hand-foot syndrome symptoms appear and continuing until the end of capecitabine therapy in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Arm A: Prior to Initiation of Capecitabine | Arm B: After Hand-foot Syndrome (HFS) Symptoms Appear
Started | 12 | 12
Started Capecitabine | 11 | 11
Completed | 10 | 7
Not Completed | 2 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — No HFS / Never Started Patch/ | 0 | 4
Not completed — Never began capecitabine | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Prior to Initiation of Capecitabine | Arm B: After Hand-foot Syndrome Symptoms Appear | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Customized [Count of Participants; unit: Participants]
  30-39 years old | 1 | 1 | 2
  40-49 years old | 4 | 4 | 8
  50-59 years old | 2 | 0 | 2
  60-69 years old | 5 | 5 | 10
  70-79 years old | 0 | 1 | 1
  80-89 years old | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 12 | 24
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 11 | 12 | 23
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 2 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 7 | 10 | 17
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Developed Hand-foot Syndrome (HFS) by Toxicity Grade
Description: Incidence and severity of hand-foot syndrome (HFS) developed during chemotherapy will be defined by using the grading system for HFS per the NCI Cancer Therapy Evaluation Program Common Terminology Criteria for Adverse Events (NCI CTCAE) version 3.0 for all patients assigned who received at least 1 cycle of capecitabine.
Time Frame: up to 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Prior to Initiation of Capecitabine | Arm B: After Hand-foot Syndrome Symptoms Appear
Number analyzed (Participants) | 11 | 11
Participants
  Grade 1 HFS | 5 | 1
  Grade 2 HFS | 5 | 6
  Grade 3 HFS | 0 | 1

2. Secondary Outcome: Frequency of Side Effects of the Transdermal Nicotine Patch
Description: Beginning from first capecitabine cycle following first use of nicotine patch up through final study visit after approximately 15 weeks of nicotine patch use. All toxicities will be graded and classified according to NCI CTCAE version 3.0.
Time Frame: Up to 15 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Prior to Initiation of Capecitabine | Arm B: After Hand-foot Syndrome Symptoms Appear
Number analyzed (Participants) | 10 | 7
Participants
  Grade 1 Nausea | 4 | 5
  Grade 1 Diarrhea | 2 | 2
  Grade 2 Diarrhea | 1 | 0
  Grade 1 Headache | 2 | 2
  Grade 3 Headache | 0 | 1
  Grade 1 Dizziness | 1 | 2
  Grade 2 Dizziness | 1 | 0
  Grade 1 Sleep Disturbance | 1 | 2
  Grade 2 Sleep Disturbance | 1 | 0
  Grade 1 Rash (at patch site) | 2 | 2
  Grade 1 Constipation | 0 | 1
  Grade 1 Stomach Pain | 0 | 1
  Grade 1 Irritability | 1 | 1
  Grade 1 Myalgia | 2 | 1
  Grade 1 Taste alteration | 1 | 1

3. Secondary Outcome: Compliance in Using the Transdermal Nicotine Patch as Measured by Patient Diary
Description: Self-report diaries of patch use beginning from capecitabine cycle following first use of nicotine patch use up through 15 weeks of possible nicotine patch use. Compliance will be reported by category (Compliant, Not Compliant, No Diaries Returned)
Time Frame: up to 15 weeks
Population: Only 2 patients returned the self-reported medication diaries
Measure: Number; unit: participants
Arm/Group | Arm A: Prior to Initiation of Capecitabine | Arm B: After Hand-foot Syndrome Symptoms Appear
Number analyzed (Participants) | 11 | 11
participants
  Compliant | 1 | 1
  Not Compliant | 0 | 0
  No Diaries Returned | 10 | 10

4. Secondary Outcome: Number of Patients Requiring Dose Reduction of Capecitabine
Description: Determined by the number of patients who required a toxicity-related, dose reduction of capecitabine during active treatment at each cycle where a dose reduction occurred.
Time Frame: up to 24 weeks
Population: No toxicities for dose reduction assessed at cycle 1. The maximum number of cycles where a dose reduction occurred was 8 for Arm A, and 5 for Arm B.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Prior to Initiation of Capecitabine | Arm B: After Hand-foot Syndrome Symptoms Appear
Number analyzed (Participants) | 11 | 11
Participants
  Treatment Cycle 2 | 3 | 4
  Treatment Cycle 3 | 3 | 5
  Treatment Cycle 4 | 0 | 1
  Treatment Cycle 5 | 1 | 1
  Treatment Cycle 6 | 0 | NA — Maximum number of cycles where a dose reduction occurred was 5 for Arm B.
  Treatment Cycle 7 | 1 | NA — Maximum number of cycles where a dose reduction occurred was 5 for Arm B.
  Treatment Cycle 8 | 1 | NA — Maximum number of cycles where a dose reduction occurred was 5 for Arm B.

5. Secondary Outcome: Number of Patients With Reported Use of Pain Medication for HFS
Description: Determine the number of patients requiring pain medication for the management of symptomatic HFS
Time Frame: Until last dose of capecitabine treatment or HFS has resolved, approximately 1 year
Measure: Count of Participants; unit: Participants
Groups:
- Arm A: Patients apply a transdermal nicotine patch once every 24 hours beginning 1 day prior to initiation of capecitabine and continuing until the end of capecitabine therapy in the absence of disease progression or unacceptable toxicity.
- Arm B: Patients apply a transdermal nicotine patch once every 24 hours beginning with the course of chemotherapy initiated after hand-foot syndrome symptoms appear and continuing until the end of capecitabine therapy in the absence of disease progression or unacceptable toxicity.
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 10 | 7
Participants | 6 | 7

6. Secondary Outcome: Number of Patients With Reported Use of Other Symptomatic Treatments for HFS
Description: Determine the number of patients utilizing additional treatments for symptomatic HFS. Additional treatments may include moisturizers, ice, and/or cooling packs
Time Frame: Until last dose of capecitabine treatment or HFS has resolved, approximately 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Prior to Initiation of Capecitabine | Arm B: After Hand-foot Syndrome Symptoms Appear
Number analyzed (Participants) | 10 | 7
Participants | 5 | 7

7. Secondary Outcome: Quality of Life as Measured by FACT-B Scale
Description: The Functional Assessment of Cancer Therapy - Breast (FACT-B) scale is widely used to measure health-related quality of life in cancer patients. The FACT-B is a 44-item self-report instrument designed to measure multidimensional quality of life (QL) in patients with breast cancer, given at screening, week 9, and week 15 assessments during nicotine patch use.
Time Frame: Up to 15 weeks
Population: Data for this endpoint was not collected
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after patient's last dose of capecitabine, approximately 1 year
Arm/Group | Arm A: Prior to Initiation of Capecitabine | Arm B: After Hand-foot Syndrome Symptoms Appear
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 8/11 | 8/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Prior to Initiation of Capecitabine (N=11) | Arm B: After Hand-foot Syndrome Symptoms Appear (N=11)
Nausea (Gastrointestinal disorders) | 4 | 8
Diarrhea (Gastrointestinal disorders) | 3 | 8
Headache (Nervous system disorders) | 2 | 4
Sleep Disturbance (Nervous system disorders) | 2 | 2
Rash (at patch site) (Injury, poisoning and procedural complications) | 2 | 2
Irritability (General disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Taste alteration (Gastrointestinal disorders) | 1 | 1
Dizziness (Nervous system disorders) | 2 | 2
Stomach Pain (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1
Mucositis (Gastrointestinal disorders) | 0 | 2
Oral ulcerations (Gastrointestinal disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study terminated earlier than expected due to low accrual

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes